CLINICAL TRIAL: NCT02558114
Title: Randomized Study of Two Treatment Strategies With Ribavirin for Chronic Hepatitis E and Severe Acute Forms
Brief Title: Ribavirin for Severe Acute and Chronic Hepatitis E Virus Infection.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RACHE
Record Dates: First submitted 2015-09-18; First posted 2015-09-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis E
MeSH Terms: conditions — Hepatitis E | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Patients will receive ribavirin during 12 weeks
  Interventions: Drug: Ribavirin
- Group B (Other): Patients will receive:
  * ribavirin during 12 weeks if RNA (Ribonucleic acid) Hepatitis E virus (HEV) is undetectable at week 4 after treatment start (adjust to renal function)
  * - ribavirin during 24 weeks if RNA (Ribonucleic acid) Hepatitis E virus (HEV) is detectable at week 4 after treatment start (adjust to renal function)
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin

SUMMARY:
The purpose of the study is to compare the efficacy, safety and recurrence rate of two therapeutic strategies with ribavirin in patients with chronic hepatitis E and severe acute hepatitis E: fixed duration of treatment for 12 weeks vs variable duration depending on the viremia within 4 weeks of the start of treatment (12 vs 24 weeks).

The purpose of the study is also improve the safety of treatment with Ribavirin by optimizing dose adjusted to renal function, plasma levels of drug and hemoglobin.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years.
* To comply with any of the following diagnoses:
* chronic Hepatitis E: HEV RNA detectable in patients with elevated transaminase levels for at least 6 months and / or HEV RNA detectable in two separated determinations by an interval of six months .
* severe acute Hepatitis E: alanine aminotransferase (ALT) levels greater than 10 times the normal limit, with HEV RNA positive, and signs of acute liver injury (International normalized ratio(INR> 1.5)); or with extrahepatic manifestations or liver failure in patients with previous liver disease.
* Signed informed consent

Exclusion Criteria:

* Terminal illness with a expected life expectancy of less than 6 months
* Patients with contraindications for treatment with Ribavirin:
* pregnancy or lactation.
* Severe hepatic impairment or decompensated cirrhosis.
* hemoglobinopathies (thalassemia, sickle cell anemia).
* history of severe pre-existing cardiac disease, including unstable heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Sustained virological response measured by HEV RNA | 48 weeks
  HEV RNA undetectable at 48 weeks after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari vall d'Hebron, Barcelona, Spain